CLINICAL TRIAL: NCT06363448
Title: Yamani Technique Versus Proline Mesh for Intraocular Lens Scleral Fixation in Aphakia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elshimaa A.Mateen, Assisstant Professor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-24-3-04PD
Record Dates: First submitted 2024-04-03; First posted 2024-04-12 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Aphakia, Postcataract
MeSH Terms: conditions — Aphakia, Postcataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yamani technique (Active Comparator): Yamani technique for aphakia
  Interventions: Procedure: Yamani Technique versus Prolene Mesh for Intraocular Lens Scleral Fixation in Aphakia
- Proline mesh for aphakia (Active Comparator): Proline mesh for aphakia
  Interventions: Procedure: Yamani Technique versus Prolene Mesh for Intraocular Lens Scleral Fixation in Aphakia

INTERVENTIONS:
Procedure: Yamani Technique versus Prolene Mesh for Intraocular Lens Scleral Fixation in Aphakia — Patients were divided into two groups to undergo classic ab externo two-point scleral fixation or flanged haptics as described by Yamani or the 2*2 proline mesh technique.

SUMMARY:
The study aims to describe a new method of sulcus fixation of intraocular lenses (IOLs) using a prolene mesh and to compare its outcomes with Yamani technique.

DETAILED DESCRIPTION:
Properly positioned posterior chamber IOL (PCIOL) offers many advantages over an anterior chamber IOL (ACIOL). The potential advantages of PCIOLs over ACIOLs include a reduction in the number of optical aberrations (e.g. magnification, aniseikonia, lens edge glare, flutter), a decreased incidence of secondary glaucoma, and free movement of the pupil to control the amount of light entering the eye.

The risk for corneal decompensation, secondary glaucoma, and cystoid macular edema may be less with PCIOLs than with ACIOLs. In the absence of capsular support, many techniques have been described to secure the haptics to the sulcus region.

All described techniques focus on IOL haptics fixation to the scleral wall at two or more points. These techniques are not free of complications, including IOL tilt, misalignment, myopic shift, IOL suture rupture, and dislocation. In a previous study, Othman et al compared classic ab-externo two-point IOL fixation with a new technique of IOL scleral fixation based on fashioning trans-scleral, a double rectangular suture sulcus reconstruction (DRSSR) to support the IOL optic, thus providing a cushion to the IOL being positioned in the sulcus.

Aim of

ELIGIBILITY:
Inclusion Criteria:

* patients aged 40 years
* aphakic patients (post-traumatic or after complicated cataract surgery without capsular support).

Exclusion Criteria:

* Corneal decompensation.
* Jeopardized specular microscopy
* retinal or choroidal detachment
* retained Intraocular foreign body
* uveitis, Scleromalacia
* Reubeosis irides
* previous anti-glaucoma surgery.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) in LogMAR | 6 months
  Best corrected visual acuity (BCVA) in LogMAR

CONTACTS AND LOCATIONS:
Overall Officials: Elshimaa A.Mateen, Doctor, Principal Investigator — Assistant professor of ophthalmology, Sohag University
Locations (2):
- Egypt (2):
  - Ophthalmology department, Sohag University, Sohag
  - Elshimaa A.Mateen, Sohag

IPD SHARING:
Plan to Share IPD: No